CLINICAL TRIAL: NCT02966496
Title: Safety and Efficacy of Implantation of Two Multifocal Intraocular Lenses in the Treatment of Senile Cataract: a Randomized Controlled Clinical Trial
Brief Title: Safety and Efficacy of Implantation of Two Multifocal Intraocular Lenses in the Treatment of Senile Cataract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qinghai University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QinghaiUH_005
Record Dates: First submitted 2016-11-09; First posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Senile Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the test group (Experimental): The patients aged 50-80 years will be randomly assigned to implantation of Acri.LISA366D multifocal aspheric IOLs in the test group.
  Interventions: Biological: Acri.LISA366D multifocal aspheric IOLs
- the control group (Experimental): The patients aged 50-80 years will be randomly assigned to implantation of TecnisZ9001 multifocal aspheric IOLs in the control group.
  Interventions: Biological: TecnisZ9001 multifocal aspheric IOLs

INTERVENTIONS:
Biological: Acri.LISA366D multifocal aspheric IOLs — The implantation of Acri.LISA366D multifocal aspheric IOLs are used in the test group.
  Arms: the test group
Biological: TecnisZ9001 multifocal aspheric IOLs — The implantation of TecnisZ9001 multifocal aspheric IOLs are used in the test group.
  Arms: the control group

SUMMARY:
This trial is designed to compare the biocompatibility and long-term visual outcomes of the Tecnis Z9001 and Acri.LISA 366D multifocal IOLs used for the treatment of senile cataract. The aim is to provide a safer biomaterial for senile cataract treatment, achieving better postoperative visual quality and fewer complications.

DETAILED DESCRIPTION:
History and current studies Aging-induced degenerative diseases are the leading cause of senile cataract. Phacoemulsification with intraocular lens (IOL) implantation is a commonly employed surgical technique for the treatment of cataract. A traditional IOL is spherical and monofocal. Traditional monofocal IOL implantation allows cataract patients to obtain good postoperative distance vision but loss of accommodation results in poor near vision. Following monofocal IOL implantation, most patients still require the use of glasses. Fortunately, the presence of multifocal IOLs solves this problem. Studies have shown that aspheric IOLs with zero or negative spherical aberration can eliminate or reduce the spherical aberration of the whole eye and can improve contrast sensitivity and night vision compared with a spherical IOL.

As first reported in 1987 by Keatea et al., multifocal IOLs were introduced to provide improved visual acuity, thus eliminating the need to wear glasses and improving the patient's quality of life. Increasing evidence-based medicine evidences have shown that multifocal IOLs are more adept to improving near vision than single-focus IOLs. To date, various types of multifocal IOLs have been developed and according to different design principles, clinically used multifocal IOLs have been divided into refraction type, diffraction type and refraction/diffraction type. Introduced in 2002, the Tecnis Z9001 diffractive multifocal aspherical IOL (Abbott Medical Optics, CA, USA) is clinically proven to give patients improved contrast vision and visual quality when compared with the common IOL, although deficiencies include postoperative glare and reduced contrast sensitivity. Emerging designs for multifocal IOLs aim to provide improvements in postoperative visual quality. The Acri.LISA 366D multifocal aspheric IOL is a relatively novel refractive/diffractive multifocal IOL that is different from traditional IOLs. Its unique optical design improves the patient's full vision and reduces the incidence of light scattering, glare and halo, which is expected to deliver better clinical outcomes. However, its long-term clinical performance and the potential incidence of complications still need further evaluation.

It is worth noting that as age increases, the increase in presbyopia, aberrations and lens scattering reduces the compensation for corneal aberrations, thereby resulting in a decrease in visual acuity and contrast sensitivity. Given this, ideal IOLs should have good biocompatibility and good resolution with no spherical aberration.

Data collection, management, analysis, and open access Data collection Clinical data will be collected and managed using an electronic data capture system. All data relevant to the trial will be recorded in electronic case report forms that will be provided by the sponsor personnel. The case report will be completed after the interview.

Data management After completion of follow-up and data confirmation, only the project manager will lock the database. The locked data will be unable to be altered and will be preserved for future reference by the Affiliated Hospital of Qinghai University in China.

Data analysis All data will be statistically analyzed by professional statisticians.

Open data Published data will be released at http://www.medresman.org.

Statistical analysis All data will be statistically analyzed by statisticians using SPSS v19.0 software. Normally distributed measurement data will be expressed as mean ± standard deviation, while non-normally distributed data will be expressed as quartiles and medians. Categorical variables will be expressed as counts and percentages. Two-sample t-test or Mann-Whitney U-test will be used for intergroup comparison of visual acuity and diopter. The chi-squared test or Fisher's exact test will be used for intergroup comparison of incidence of histocompatibility reactions between the implant and host tissues and the percentage of complications. A value of P < O.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as age-related cataract.
* Corneal astigmatism < 1.0 D
* Lens hardness, II-III
* Initial surgery on the eye
* Age 50-80 years
* Healthy and able to tolerate anesthesia and surgery

Exclusion Criteria:

* Glaucoma or secondary vision loss resulting from diabetes, hypertension, intracranial tumors and neurological diseases
* Fundus disease, corneal edema, corneal opacity, endophthalmitis, and/or iris adhesion.
* Prior experience of eye surgery
* Failure to make regular referrals
* Autoimmune disease, mental illness or other serious systemic disease
* Inability to cooperate with the researchers
* Inability to tolerate surgery
* Sensitivity, anxiety or the pursuit of perfection
* Inability to give informed consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of cataract participants with good biocompatibility of intraocular lens implants | month 12 after surgery
  Good engraftment, epithelialization, no neovascularization, retained transparency, no host inflammatory reaction.

SECONDARY OUTCOMES:
Visual acuity | at month 1, month 3, month 6, month 12 and month 24 after surgery
  Best spectacle corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Ping Yu, Master, Principal Investigator — Affiliated Hospital of Qinghai University

IPD SHARING:
Plan to Share IPD: Undecided